CLINICAL TRIAL: NCT01347645
Title: An Open-Label, Multicenter, Randomized Phase Ib/II Study of Irinotecan Plus E7820 Versus FOLFIRI in Second-Line Therapy in Patients With Locally Advanced or Metastatic Colon or Rectal Cancer
Brief Title: Irinotecan Plus E7820 Versus FOLFIRI in Second-Line Therapy in Patients With Locally Advanced or Metastatic Colon or Rectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor due to E7820 plus irinotecan being potentially inferior to FOLFIRI
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7820-702; 2011-001762-18 (EudraCT Number)
Record Dates: First submitted 2011-04-28; First posted 2011-05-04 (Estimated); Results first posted 2022-11-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: locally advanced; metastatic colon; rectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — IFL protocol; N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Experimental Irinotecan plus E7820
  Interventions: Drug: E7820
- 2 (Active Comparator): FOLFIRI alone
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFIRI — Comparator dose and mode of administration The FOLFIRI regimen consists of irinotecan at 180 mg/m2 (IV infusion) on Day 1 of each 14-day cycle, leucovorin at 200 mg/m2 (400 mg/m2 if using d,l-racemic mixture of leucovorin) by IV infusion on Day 1 of each cycle, and 5-FU at 400 mg/m2 as an IV bolus injection followed by a total of 2400 mg/m2 by continuous IV infusion over 46 hours over Days 1 and 2 via an ambulatory programmable pump (the use of an ambulatory pump is optional).
  Arms: 2
Drug: E7820 — Test product: dose and mode of administration:
  E7820 is administered orally in tablet form once daily, every day of each 14-day treatment cycle. For the Phase Ib portion, the doses will be 40 mg/day, 70 mg/day, and 100 mg/day, and for the Pase II portion, the dose will be the MTD in combination with Irinotecan, as determined during the Phase ib portion of the study.
  The irinotecan regimen consists of an irinotecan dose of 180 mg/m2 by IV infusion once every 2 weeks (Day 1 of each 14-day cycle).
  Arms: 1

SUMMARY:
The purpose of the Phase Ib portion is to find out the highest dose of study drug that can safely be given when tested in a small group of subjects.

The purpose of the Phase II portion is to find out how safe the study drug is when taken at the highest dose in a larger group of subjects.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of a Phase Ib portion: a safety run-in period with 3 ascending doses of E7820; and a Phase II portion: a randomized 2-arm design. Approximately 95 patients with measurable, nonresectable locally advanced or metastatic colorectal adenocarcinoma, who have failed first-line chemotherapy, will be enrolled in the study (approximately 12 to 15 patients in the Phase Ib portion and 80 patients in the Phase II portion). Patients will only participate in either the Phase Ib or the Phase II portion of the study. Patients will receive up to a planned total of 12 cycles of study treatment unless there is occurrence of progressive disease, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurs first. After 12 cycles, patients who demonstrate clinical benefit may continue single agent E7820 for long as clinical benefit is sustained and the treatment is well tolerated. If the treating physician does not feel comfortable discontinuing chemotherapy after 12 cycles, further chemotherapy may be considered following discussion with the medical monitor and sponsor.

ELIGIBILITY:
Inclusion Criteria:

Patients may be entered in the study only if they meet all of the following criteria:

1. Male or female patient greater than or equal to 18 years of age;
2. Histologically or cytologically confirmed nonresectable locally advanced or metastatic colorectal adenocarcinoma;
3. Patients must have failed a first-line chemotherapy regimen for nonresectable locally advanced or mCRC (first-line 5-FU-based therapies, including but not limited to FOLFOX, FOLFOX 4, mFOLFOX6, CapeOX, single-agent capecitabine, infusional 5-FU, or other chemotherapies. Bevacizumab, cetuximab, panitumumab, and EGFR inhibitors are allowed. Prior treatment with irinotecan or FOLFIRI is not allowed for Phase II). For Phase Ib only, up to 3 prior therapies are allowed (including non-irinotecan containing therapies and adjuvant therapy);
4. At least 1 site of measurable disease by the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) criteria;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of less than or equal to 2;
6. Patients must have adequate renal function as evidenced by serum creatinine less than 2 mg/dL and creatinine clearance greater than 50 mL/minute per the Cockcroft and Gault formula;
7. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, platelets greater than100 x 109/L, hemoglobin greater than or equal to 9.0 g/dL (a hemoglobin less than 9.0 g/dL at Screening is acceptable if it is corrected to greater than or equal to 9 g/dL by growth factor or transfusion prior to the first dose);
8. Patients must have adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limit of the normal range (ULN), and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 X ULN (in the case of liver metastases, less than or equal to 5 X ULN).If there are bone metastases, liver-specific alkaline phosphatase may be separated from the total and used to assess liver function instead of total alkaline phosphatase;
9. For patients with hypertension, it must be well controlled. If a patient presents with poorly controlled hypertension, defined as a mean systolic blood pressure greater than or equal to140 mm Hg or mean diastolic blood pressure greater than or equal to 90 mm Hg,antihypertensive medication(s) should be initiated or adjusted with a goal to control the blood pressure less than 140/90 mm Hg. Blood pressure must be reassessed on 2 occasions, consecutively, that are separated by a minimum of 24 hours;
10. Male or female patients of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment;
11. Females of childbearing potential must have a negative serum pregnancy test at Screening;
12. Females may not be breastfeeding; Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

1. Received chemotherapy, targeted therapy, radiotherapy, surgery, immunotherapy, or treatment in another clinical study within the 30 days prior to commencing study treatment or have not recovered from side effects of all treatment-related toxicities to Grade less than or equal to 1, except for peripheral neuropathy (Grade 1 and Grade 2 are permitted) and alopecia;
2. Previously received irinotecan or irinotecan derivatives in Phase II (irinotecan-containing regimens are allowed in Phase Ib);
3. Previously received anti-alpha 2 integrin therapy;
4. History of other malignancies except: (1) adequately treated basal or squamous cell carcinoma of the skin; (2) curatively treated in situ carcinoma of the uterine cervix; or (3) other curatively treated solid tumor with no evidence of disease for greater than or equal to 5 years;
5. Presence of brain metastases, unless the patient has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
6. Are currently receiving any other anticancer treatment;
7. Serious non-healing wound, ulcer, or active bone fracture;
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for a major surgical procedure during the course of the study;
9. Refractory nausea and vomiting, malabsorption, significant bowel resection, or any other medical condition that would preclude adequate absorption or result in the inability to take oral medication;
10. Significant cardiovascular impairment (history of congestive heart failure New York Heart Association [NYHA] Grade greater than 2, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
11. Active hemoptysis (defined as bright red blood of 1/2 teaspoon or more) within the 30 days prior to study entry;
12. Current or recent use (within 7 days) of full-dose warfarin (except low-dose warfarin as required to maintain patency of pre-existing, permanent indwelling IV catheters). For patients receiving warfarin, International Normalization Ratio (INR) should be less than 1.5. Patients may have prophylactic use of low molecular weight heparin; however, therapeutic use of heparin or low molecular weight heparin is not acceptable;
13. History of bleeding diathesis or coagulopathy;
14. Any history of cerebral vascular accident, transient ischemic attack, or Grade greater than or equal to 2 peripheral vascular disease, unless they have had no evidence of active disease for at least 6 months prior to randomization;
15. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1, unless affected area has been removed surgically;
16. Patients with organ allografts requiring immunosuppression;
17. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or active hepatitis C positive;
18. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan, 5-FU, or leucovorin;
19. Hypersensitivity to sulfonamide derivatives;
20. Have any medical condition that would interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, Study Director — Quintiles, Inc.
Locations (36):
- United States (6):
  - Birmingham, Alabama
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Ann Arbor, Michigan
  - Berkeley Heights, New Jersey
  - Bismarck, North Dakota
- Argentina (4):
  - Ciudad Autonoma de Buenos Aires, Buenos Aires
  - La Rioja, LA Rioha
  - Rosario, Santa Fe Province
  - Córdoba
- Australia (11):
  - Coffs Harbour, New South Wales
  - Concord, New South Wales
  - Townsville, Queensland
  - Elizabeth Vale, South Australia
  - Kurralta Park, South Australia
  - Woodville South, South Australia
  - Carlton, Victoria
  - Clayton, Victoria
  - Epping, Victoria
  - Frankston, Victoria
  - Wodonga, Victoria
- Brazil (7):
  - Belo Horizonte, Minas Gerais
  - Novo Hamburgo, Rio Grande do Sul
  - Passo Fundo, Rio Grande do Sul
  - Port Alegre, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Jaú, São Paulo
  - Rio de Janeiro
- Russia (5):
  - Arkhangelsk
  - Chelyabinsk
  - Moscow
  - Saint Petersburg
  - Sochi
- Ukraine (3):
  - Dnipropetrovsk
  - Kharkiv
  - Uzhhorod

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 investigative sites in Argentina, Australia, Brazil, Russian Federation, Ukraine, and the United States from 30 September 2011 to 22 June 2015.
Pre-assignment Details: A total of 82 participants were enrolled in this study. This study consisted of two phases: Phase 1b and Phase 2. In Phase 1b, 14 participants were enrolled and received study treatment and in Phase 2, 68 participants were enrolled and received the study treatment. Participants were randomized in a 1:1 ratio and received either E7820 in combination with irinotecan or FOLFIRI.
Groups:
- Phase 1b: Cohort 1: E7820 40 mg + Irinotecan: Participants received E7820 40 milligram (mg) tablets, orally, once daily of each 14-day treatment cycle in combination with irinotecan 180 milligram per square meter (mg/m^2) as an intravenous infusion on Day 1 of each 14-day cycle (once every 2 weeks) for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until disease progression (PD), unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 2: E7820 70 mg + Irinotecan: Participants received E7820 70 mg tablets, orally, once daily of each 14-day treatment cycle in combination with irinotecan 180 mg/m^2 as an intravenous infusion on Day 1 of each 14-day cycle (once every 2 weeks) for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 3: E7820 100 mg + Irinotecan: Participants received E7820 100 mg tablets, orally, once daily of each 14-day treatment cycle in combination with irinotecan 180 mg/m^2 as an intravenous infusion on Day 1 of each 14-day cycle (once every 2 weeks) for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 2: E7820 70 mg + Irinotecan: Participants received E7820 70 mg (changed to 50 mg as per protocol amendment 06) as Recommended Phase 2 dose (RP2D) tablets, orally, once daily of each 14-day treatment cycle on Day 1 with Irinotecan 180 mg/m^2 as an intravenous infusion on Day 1 of each 14-day cycle for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 2: Folfiri: Participants received the FOLFIRI regimen, which consisted of irinotecan at 180 mg/m^2 as an intravenous infusion and leucovorin at 200 mg/m^2 by intravenous infusion on Day 1 of each cycle, and 5-FU at 400 mg/m^2 as an intravenous bolus injection followed by a total of 2400 mg/m^2 by continuous IV infusion over 46 hours over Days 1 and 2 via infusion for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Period: Overall Study
Arm/Group | Phase 1b: Cohort 1: E7820 40 mg + Irinotecan | Phase 1b: Cohort 2: E7820 70 mg + Irinotecan | Phase 1b: Cohort 3: E7820 100 mg + Irinotecan | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Started | 3 | 8 | 3 | 34 | 34
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 3 | 34 | 34
Not completed — Death | 1 | 5 | 2 | 7 | 7
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 1
Not completed — Study termination by Sponsor due to E7820 plus irinotecan being potentially inferior to FOLFIRI | 0 | 2 | 1 | 22 | 20
Not completed — Other | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all the participants who received at least one dose of study drug and who had at least one safety assessment following the first dose.
Groups:
- Phase 1b: Cohort 1: E7820 40 mg + Irinotecan: Participants received E7820 40 mg tablets, orally, once daily of each 14-day treatment cycle in combination with irinotecan 180 milligram per square meter (mg/m^2) as an intravenous infusion on Day 1 of each 14-day cycle (once every 2 weeks) for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1: E7820 40 mg + Irinotecan | Phase 1b: Cohort 2: E7820 70 mg + Irinotecan | Phase 1b: Cohort 3: E7820 100 mg + Irinotecan | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri | Total
Number analyzed (Participants) | 3 | 8 | 3 | 34 | 34 | 82
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 85 years | 3 | 8 | 3 | 34 | 34 | 82
  >=85 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 19 | 16 | 40
  Male | 2 | 5 | 2 | 15 | 18 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) of E7820 With Irinotecan as Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0
Description: MTD: maximum dose that was determined to be safe and tolerable for Phase 2.If two dose limiting toxicities (DLTs) occurred at any dose level,MTD: preceding dose/intermediate dose.DLT was graded according to CTCAE v4.0. Includes >= Grade 3(G3) peripheral neuropathy,>=G3 nausea/vomiting despite optimal anti-emetic treatment, any other non-hematologic toxicity of >=G3(except alopecia, single abnormal laboratory values Investigator judged unlikely related to study therapy, had no clinical correlate, resolved in 7 days, hypersensitivity reaction to any of compounds),Grade 4 neutropenia lasting over 7 days,febrile neutropenia(defined as fever >=38.5 degrees Celsius with absolute neutrophil count below 1.0*10^9 per liter, G3 thrombocytopenia with nontraumatic bleeding(without therapeutic systemic anticoagulation)requiring platelet transfusion,Grade 4 thrombocytopenia (with/without nontraumatic bleeding),any study drug-related death,other toxicity dose escalation committee believed to be DLT.
Time Frame: Up to 12 cycles (each cycle length =14 days)
Population: The safety population included all the participants enrolled in the Phase 1b portion of this study, except for those who (i) dropped out of the study prior to receiving any study drug, or (ii) were without any safety assessment following the first dose of study drug.
Measure: Number; unit: milligram (mg)
Groups:
- Phase 1b, All Participants: Participants received E7820 40 mg, 70 mg and 100 mg tablets, orally, once daily of each 14-day treatment cycle in combination with irinotecan 180 mg/m^2 as an intravenous infusion on Day 1 of each 14-day cycle (once every 2 weeks) for up to 12 cycles. After 12 cycles, at the discretion of the Investigator and in consultation with the Medical Monitor, participants who were experiencing clinical benefit continued their assigned treatment until PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Arm/Group | Phase 1b, All Participants
Number analyzed (Participants) | 14
milligram (mg) | NA — The MTD for E7820 in combination with irinotecan was not determined. Based on dose reductions and interruptions at the 100 mg dose, it was decided that the E7820 Phase 2 dose would be 70 mg once daily.

2. Primary Outcome: Phase 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE is defined as an adverse event that had an onset date, or a worsening in severity on or after the first dose of study drug up to the end of the study. Number of participants with TEAEs are reported based on safety assessments of laboratory tests, physical examination, examining bowel movements, regular measurement of vital signs, eastern cooperative oncology group-performance status and electrocardiogram parameter values. SAE is any untoward medical occurrence that at any dose: resulted in death; life threatening required inpatient hospitalization; resulted in persistent, significant disability; is congenital anomaly/birth defect or medically important due to other reasons than above mentioned criteria. Number of participants with TEAEs and SAEs were reported.
Time Frame: From the first dose of study drug up to 28 days after last dose (Up to 1 year and 3 months)
Population: The safety population included all participants enrolled and randomized to treatment in the Phase 2 portion of this study, except for those who (i) dropped out prior to receiving any study drug, or (ii) were without any safety assessment following the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Number analyzed (Participants) | 34 | 34
Participants
  TEAEs | 34 | 34
  SAEs | 10 | 8

3. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization of a participant until the sooner of (1) the date of first documented progression of such participant's disease (PD) based on Investigator assessments according to response evaluation criteria in solid tumor (RECIST) version (v) 1.1. or; (2) the date of such participant's death due to any cause. PD is defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From date of randomization up to 1 year and 2 months
Population: Modified intent-to-treat (MITT) analysis set included all participants who were randomized and received at least one dose of study medication without major protocol eligibility violations.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Number analyzed (Participants) | 34 | 34
weeks | 17.1 [9.00 to 32.29] | 33.7 [24.14 to 45.43]

4. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as time from the date of randomization of a participant until the date of death of such participant, regardless of the actual cause of the participant's death.
Time Frame: From date of randomization up to 1 year and 2 months
Population: MITT analysis set included all participants who were randomized and received at least one dose of study medication without major protocol eligibility violations.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Number analyzed (Participants) | 34 | 34
weeks | NA [NA to NA] — Overall survival could not be estimated due to insufficient number of participants reached the event during the study. | NA [NA to NA] — Overall survival could not be estimated due to insufficient number of participants reached the event during the study.

5. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP is defined as time from the date of randomization of a participant until the date of first documented progression of such participant's disease. PD is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking in reference the smallest summed longest diameters on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. The appearance of 1 or more new lesions was also considered progression.
Time Frame: From date of randomization up to 1 year and 2 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Number analyzed (Participants) | 34 | 34
weeks | 23.7 [14.43 to 33.00] | 33.7 [24.14 to 45.43]

6. Secondary Outcome: Phase 2: Percentage of Participants With Overall Response
Description: ORR is defined as percentage of participants in the study whose best overall response is either complete response (CR) or partial response (PR) based on RECIST v1.1. CR is defined as complete disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to less than 10 mm. PR is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline summed longest diameters.
Time Frame: From date of randomization up to 1 year and 2 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
Number analyzed (Participants) | 34 | 34
percentage of participants | 20.6 [8.7 to 37.9] | 20.6 [8.7 to 37.9]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 28 days after last dose (Up to 1 year and 3 months)
Arm/Group | Phase 1b: Cohort 1: E7820 40 mg + Irinotecan | Phase 1b: Cohort 2: E7820 70 mg + Irinotecan | Phase 1b: Cohort 3: E7820 100 mg + Irinotecan | Phase 2: E7820 70 mg + Irinotecan | Phase 2: Folfiri
All-Cause Mortality (participants affected / at risk) | 1/3 | 5/8 | 2/3 | 7/34 | 7/34
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/8 | 0/3 | 10/34 | 8/34
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 3/3 | 33/34 | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: E7820 40 mg + Irinotecan (N=3) | Phase 1b: Cohort 2: E7820 70 mg + Irinotecan (N=8) | Phase 1b: Cohort 3: E7820 100 mg + Irinotecan (N=3) | Phase 2: E7820 70 mg + Irinotecan (N=34) | Phase 2: Folfiri (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: E7820 40 mg + Irinotecan (N=3) | Phase 1b: Cohort 2: E7820 70 mg + Irinotecan (N=8) | Phase 1b: Cohort 3: E7820 100 mg + Irinotecan (N=3) | Phase 2: E7820 70 mg + Irinotecan (N=34) | Phase 2: Folfiri (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 2 (4) | 11 (25) | 8 (19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (8) | 0 (0) | 10 (49) | 8 (19)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (18) | 1 (5) | 19 (81) | 19 (52)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 1 (1) | 2 (9) | 5 (6) | 6 (13)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 4 (10) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (20) | 6 (9) | 3 (9) | 16 (45) | 14 (49)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (23) | 4 (4) | 2 (3) | 9 (18) | 16 (58)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (9) | 3 (3) | 9 (22)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 6 (9) | 9 (19)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (18) | 5 (6) | 2 (2) | 7 (11) | 9 (12)
Generalised oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (5) | 1 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 4 (5) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (7) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (3) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 2 (6) | 1 (1) | 0 (0) | 3 (4) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 16 (20) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes